CLINICAL TRIAL: NCT04146116
Title: Feasibility of Pre-operative Povidone Iodine Decolonization Among Orthopedic Trauma Surgery Patients To Reduce Staphylococcus Aureus Surgical Site Infections
Brief Title: Nasal Decolonization for Orthopedic Trauma Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: Professional Disposables International, Inc. (Industry)
Responsible Party: Principal Investigator, Marin L. Schweizer, PhD, Associate Professor, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 201812801
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Results first posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Surgical Site Infection
Keywords: nasal decolonization; Orthopedic trauma surgery
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: 50 patients will receive PROFEND intranasal povidone-iodine prior to surgery and after surgery. The study aims to evaluate the real-world effectiveness of PROFEND® in reducing S. aureus colonization and surgical site infections (SSIs).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Nasal povidone-iodine (Experimental): Intranasal povidone-iodine (PDI PROFEND) will be applied to the patients' noses before orthopedic trauma surgery and after surgery. This intranasal povidone-iodine was developed under the Tentative Final Monograph for Health-Care Antiseptic Drug Products 21 CFR Parts 333 and 369 (Docket # 75N-183H), Federal Register Volume 59, Number 116, Friday, June 17, 1994, Proposed Rules. However, the product need not be controlled like a pharmaceutical drug. The product may be stored and controlled similarly to an iodine or alcohol skin preparation product.
  Interventions: Drug: intranasal povidone-iodine

INTERVENTIONS:
Drug: intranasal povidone-iodine — povidone-iodine USP, 10% w/w antiseptic
  Other Names: PROFEND

SUMMARY:
Many surgical site infections are caused by bacteria that is transferred from a patient's nose to their open surgical wound. Some small studies have shown that putting povidone-iodine in a patient's nose reduces this risk. This study aims to evaluate the real-world effectiveness of nasal povidone-iodine (PROFEND®) in a group of 50 patients at the University of Iowa.

DETAILED DESCRIPTION:
Aim 1. Evaluate the real-world effectiveness of intranasal povidone-iodine (PROFEND®) in reducing Staphylococcus aureus colonization and surgical site infections (SSIs).

Aim 1a. Evaluate patients after surgery to determine S. aureus colonization and to survey patients on tolerability of intranasal povidone-iodine decolonization. The intranasal povidone-iodine swab will be administered to the patient's nares around one hour prior to the first surgical incision. It will then be re-applied around 12 hours later, for a total of two applications within a 24 hour period.

During the same visit at 24 hours after surgery, patients will also be administered a questionnaire to determine the tolerability of intranasal povidone-iodine decolonization. Questions will be asked about adverse events (e.g., itching, irritation) and how intranasal povidone-iodine felt (very pleasant, pleasant, neutral, unpleasant, very unpleasant).

Based on the data obtained from this aim, we will summarize the patient acceptance of intranasal povidone-iodine.

Aim 1b. Compare the rates of SSI among orthopaedic trauma surgery patients who received intranasal povidone-iodine to similar patients who received orthopedic trauma surgery before intranasal povidone-iodine implementation.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing operative fixation of lower extremity fractures at the University of Iowa during the study period.

Exclusion Criteria:

* Patients unable to provide informed consent due to head trauma or dementia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marin L Schweizer, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Obtained informed consent in the day of surgery area of the hospital prior to surgery.
Period: Overall Study
Arm/Group | Nasal Povidone-iodine
Started | 65
Completed | 51
Not Completed | 14

BASELINE CHARACTERISTICS:
Population: Patients who received orthopedic trauma surgery who consented to the intervention.
Arm/Group | Nasal Povidone-iodine
Number analyzed (Participants) | 51
Age, Customized [Count of Participants; unit: Participants] — Population: Not collected.
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Not collected
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Staphylococcus Aureus Nasal Colonization
Description: A dry, sterile, rayon swab will be used to sample the anterior apex portion of the right and left nostril. This swab will be tested for S. aureus bacteria. If bacteria are found in either nostril, the participant is categorized as being colonized with S. aureus (e.g. carries the bacteria in their nose with no signs or symptoms of infection).
Time Frame: Within 6 hours after first dose of povidone-iodine
Population: All patients who received 2 doses of nasal povidone-iodine (pre-surgery and post-surgery)
Measure: Count of Participants; unit: Participants
Arm/Group | Nasal Povidone-iodine
Number analyzed (Participants) | 51
Participants | 12

2. Secondary Outcome: Number of Participants With Staphylococcus Aureus Nasal Colonization
Description: A dry, sterile, rayon swab will be used to sample the anterior apex portion of the right and left nostril. This swab will be tested for S. aureus bacteria. This swab will be tested for S. aureus bacteria. If bacteria are found in either nostril, the participant is categorized as being colonized with S. aureus (e.g. carries the bacteria in their nose with no signs or symptoms of infection).
Time Frame: Within 24 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Nasal Povidone-iodine
Number analyzed (Participants) | 51
Participants | 2

3. Secondary Outcome: Number of Participants With Surgical Site Infection
Description: Surgical site infection as defined by the Centers for Disease Control and Prevention National Healthcare Safety Network.
Time Frame: Within 30 days of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Nasal Povidone-iodine
Number analyzed (Participants) | 51
Participants | 0

ADVERSE EVENTS:
Time Frame: Within 24 hours of initial application
Description: Collected via survey
Arm/Group | Nasal Povidone-iodine
All-Cause Mortality (participants affected / at risk) | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 6/51
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nasal Povidone-iodine (N=51)
Stinging in the Nose (Product Issues) | 3 (3) — Stinging in the nose assessed within 24 hours of initial application
Burning sensation (Product Issues) | 1 (1) — Burning sensation in the nose assessed within 24 hours of initial application
Sore Throat (Product Issues) | 1 (1) — Sore throat assessed within 24 hours of initial application
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Cough assessed within 24 hours of initial application

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-07-18): https://cdn.clinicaltrials.gov/large-docs/16/NCT04146116/Prot_002.pdf
  • Informed Consent Form (2019-10-16): https://cdn.clinicaltrials.gov/large-docs/16/NCT04146116/ICF_001.pdf